CLINICAL TRIAL: NCT02197676
Title: A Phase II Trial of SGI-110 in Patients With IPSS High and Int 2 Myelodysplastic Syndrome, Acute Myeloid Leukemia With 20-30% Marrow Blasts or Chronic Myelomonocytic Leukemia Type 2 Not Responding to Azacitidine or Decitabine After at Least 6 Courses or Relapsing After a Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-SGI-110
Record Dates: First submitted 2014-04-29; First posted 2014-07-23 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: MDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGI-110 (Experimental)
  Interventions: Drug: SGI-110 administration

INTERVENTIONS:
Drug: SGI-110 administration — SGI-110 will be administered SC at 60 mg/m²/day x5 consecutive days for each cycle. Cycle duration is 28 days. Patients with Complete Remission (CR), Partial Remission (PR), marrow CR or Hematological Improvement (HI) after 6 Cycles of therapy (IWG 2006 criteria) may continue treatment until progression.
  A dose reduction to 45 and even 30 mg/m²/day will be made in case of haematological toxicity. Patients with no response (NR) to treatment will be withdrawn from the protocol after the last treatment Cycle.

SUMMARY:
Treatment of patients with WHO defined IPSS int 2 and high risk MDS , AML with 20-30% marrow blasts and CMML type 2, after failure of azacitidine or decitabine exposure for at least 6 courses, or relapse after initial response.

DETAILED DESCRIPTION:
All eligible patients will be treated with SGI-110 for 9 cycles of 28 days.

Patients who meet eligibility criteria will be administered subcutaneous SGI-110 at 60mg/m²/d one time daily for 5 days. Each cycle will last 28 days with SGI-110 starting on day 1 of each cycle. Patients will receive at least 9 cycles unless overt progression is documented. (Overt progression will be defined by the presence of more than 30% marrow blasts and doubling of marrow blast percentage from onset of SGI-110). Dose reduction to 45 and even 30 mg/m²/d will be made in case of toxicity.

Patients with Complete Remission (CR), Partial Remission (PR), marrow CR, Hematological Improvement (HI) or stable disease (SD) after 6 Cycles of therapy (IWG 2006 criteria) may receive 3 additional cycles. Response will be re-evaluated after 9 cycles. Patients with no response (NR) to treatment after 9 cycles will be withdrawn from the protocol. Patients with progression at any time will be withdrawn from the protocol after the last treatment Cycle.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome including the following categories of the WHO classification: refractory anemia with excess blasts (RAEB), non-proliferative chronic myelomonocytic leukemia (CMML) (leukocytes < 13 G/L but > 10% marrow blasts), AML with 20-30% marrow blasts (RAEB-T according to the FAB classification), at screening time.
* Prior treatment with azacitidine or decitabine for at least 6 courses without response(CR, PR, marrow CR or stable disease with HI according to IWG 2006 criteria) or relapsing after a response. Non responders will be eligible only in the absence of overt progression, ie AML progression (if patients had no AML at onset of azacitidine/decitabine) or doubling of marrow blast percentage between onset of azacitidine/decitabine and screening
* IPSS score >1 (IPSS: Int-2 or High).
* Age ≥ 18 years.
* Normal liver function, defined by total bilirubin and transaminases less than 1.5 times the upper limit of normal.
* Normal renal function, defined by creatinine less than 1.5 times the upper limit of normal, creatinine clearance ≥ 50 mL/min.
* Patient is known not to be refractory to platelet transfusions.
* Written informed consent.
* Patient must understand and voluntarily sign consent form.
* Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements.
* ECOG performance status between 0-2 at the time of screening.
* Women of chilbearing potential* must:

  1. Understand the study drug is expected to have a teratogenic risk
  2. Agree to have a medically supervised pregnancy test on the day of the study visit or in the 3 days prior to the study visit once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence. The test should ensure the subject is not pregnant when she starts treatment.
  3. Agree to have a medically supervised pregnancy test every 4 weeks including 2 months after the end of study treatment, except in the case of confirmed tubal sterilization. These pregnancy tests should be performed on the day of the study visit or in the 3 days prior to the study visit. This requirement also applies to women of childbearing potential who practice complete and continued abstinence
  4. Agree to use, and to be able to comply with, Two medically acceptable contraceptive measures without interruption, 4 weeks before starting study drug throughout the entire duration study drug therapy (including doses interruptions) and for 2 months after the end of the study drug therapy even if she has amenorrhoea. This applies unless the subject commits to absolute and continuous abstinence confirmed on a monthly basis, to avoid pregnancy for the duration of study.
  5. Understand that even if she has amenorrhea, she must follow all the advice on effective contraception.
  6. She understands the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy
* Men must: Agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and for a further 2 3 months after the end of treatment if their partner is of childbearing potential.

Exclusion Criteria:

* Severe infection or any other uncontrolled severe condition.
* Significant cardiac disease - NYHA Class III or IV or having suffered a myocardial infarction in the last 6 months.
* Less than 30 days since prior treatment with growth factors (EPO, G-CSF).
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
* Active cancer, or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast.
* Patient already enrolled in another therapeutic trial of an investigational drug.
* HIV infection or active hepatitis B or C.
* Women who are or could become pregnant or who are currently breastfeeding.
* Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form.
* Patient eligible for allotransplantation.
* Known allergy to SGI-110 or any of its excipients.
* No affiliation to an insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 month
  Number of complete Remission (CR), CR with incomplete hematological recovery (CRi), Partial Remission (PR), Marrow CR and Hematological Improvement (HI) according to IWG 2006 criteria after 6 treatment cycles

SECONDARY OUTCOMES:
Duration of response | 4 years
  Measured from the date an objective response was achieved to the date of relapse or progression (cf. definition in appendix 5) or the date of last contact if no event occurred.
Adverse event | After 1 month
  Patients must have received at least one dose of treatment in order to be considered evaluable for toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fenaux, PHD, Principal Investigator — GFM; Marie Sébert, PHD, Principal Investigator — Saint-Louis Hospital, PARIS; Lionel Ades, PHD, Principal Investigator — Saint Louis hospital, Paris
Locations (27):
- France (27):
  - CH Angers, Angers
  - CH Avignon, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU Clémenceau, Caen
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - CHRU Limoges, Limoges
  - CH Lyon Sud, Lyon
  - Hôpital Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Clinique Beausoleil (Montpellier), Montpellier
  - CHU de nantes, Nantes
  - Centre Catherine de Sienne (Nantes), Nantes
  - CHU de Nice - Hopital de l'Archet 1, Nice
  - CHR Orléans, Orléans
  - Hopital St Louis T4, Paris
  - Centre Hospitalier Joffre, Perpignan
  - CHU de Haut-Lévèque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier de la région d'Annecy, Pringy
  - Centre Henri Becquerel, Rouen
  - Chu Purpan, Toulouse
  - Hopital Purpan Service d'Hématologie Clinique, Toulouse
  - CHU Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy